CLINICAL TRIAL: NCT01828229
Title: Consequences of Human Inactivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Anders Rasmussen Rinnov, Administrator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-4-2009-082
Record Dates: First submitted 2013-04-05; First posted 2013-04-10 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Inactivity; Obesity; Type 2 Diabetes
Keywords: Inactivity; Obesity; Type 2 diabetes; glucose metabolism; Lipid metabolism; Cognitive function
MeSH Terms: conditions — Sedentary Behavior; Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- female inactivity and hypercaloric diet (Experimental): inactivity and hypercaloric diet in women for two weeks
  Interventions: Behavioral: female inactivity and hypercaloric diet
- inactivity (Experimental): Inactivity for two weeks
  Interventions: Behavioral: inactivity
- inactivity and hypercaloric diet (Experimental): inactivity and hypercaloric diet for two weeks
  Interventions: Behavioral: inactivity and hypercaloric diet
- normal activity and hypercaloric diet (Experimental): Normal activity and hypercaloric diet for two weeks
  Interventions: Behavioral: normal activity and hypercaloric diet
- inactivity and iso-caloric diet (Active Comparator): inactivity and iso-caloric diet for two weeks
  Interventions: Behavioral: inactivity and iso-caloric diet

INTERVENTIONS:
Behavioral: female inactivity and hypercaloric diet — female inactivity and hypercaloric diet for 2 weeks
  Arms: female inactivity and hypercaloric diet
Behavioral: inactivity — inactivity for 2 weeks
  Arms: inactivity
Behavioral: inactivity and hypercaloric diet — inactivity and hypercaloric diet for 2 weeks
  Arms: inactivity and hypercaloric diet
Behavioral: normal activity and hypercaloric diet — normal activity and hypercaloric diet for 2 weeks
  Arms: normal activity and hypercaloric diet
Behavioral: inactivity and iso-caloric diet — inactivity and iso-caloric diet for 2 weeks
  Arms: inactivity and iso-caloric diet

SUMMARY:
Epidemiological studies as well as both longitudinal animal and human inactivity studies indicate that low physical activity is associated with the pathophysiology of type 2 diabetes mellitus (T2DM) and obesity, and recently it has been estimated that physical inactivity (worldwide) causes 7% of the burden of disease related to e.g. T2DM. Physical inactivity, a high energy dietary intake, and T2DM are also associated with dementia, depression, and impaired cognitive function. It is critical that we understand how inactivity alters body composition, glucose and lipid metabolism, and cognitive function, if normal physical activity can prevent these changes, and if there are any differences between sexes.

The present protocol is divided in several in several sub-studies:

1. To test whether and how a physically inactive lifestyle will influence body composition, glucose and lipid metabolism, and cognitive function.
2. To test whether normal physical activity can prevent the deleterious effect of a physically inactive lifestyle despite a high-caloric intake.
3. To test whether the influence of a physically inactive lifestyle combined with a high-caloric intake differs between sexes.

ELIGIBILITY:
Inclusion Criteria:

* Normal physical active
* Healthy
* 18-40 y of age
* Non-smokers

Exclusion Criteria:

* Pregnancy
* Diabetes in family

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | 2 weeks
  Area under the curve of plasma glucose and insulin levels during an oral glucose tolerance test

SECONDARY OUTCOMES:
visceral adiposity | 2 weeks
  Amount of visceral fat is determined by MRI scans

OTHER OUTCOMES:
Cognitive function | 2 weeks
  Assessed by the Conner's Continuous Performance Test II 2000
aerobic fitness | 2 weeks
  maximal oxygen uptake (VO2max) was measured during an incremental exercise test performed on a cycle ergometer

CONTACTS AND LOCATIONS:
Locations (1):
- Center og inflammation and metabolism, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Background] Olsen RH, Krogh-Madsen R, Thomsen C, Booth FW, Pedersen BK. Metabolic responses to reduced daily steps in healthy nonexercising men. JAMA. 2008 Mar 19;299(11):1261-3. doi: 10.1001/jama.299.11.1259. No abstract available. PMID 18349087
- [Result] Krogh-Madsen R, Thyfault JP, Broholm C, Mortensen OH, Olsen RH, Mounier R, Plomgaard P, van Hall G, Booth FW, Pedersen BK. A 2-wk reduction of ambulatory activity attenuates peripheral insulin sensitivity. J Appl Physiol (1985). 2010 May;108(5):1034-40. doi: 10.1152/japplphysiol.00977.2009. Epub 2009 Dec 31. PMID 20044474
- [Result] Knudsen SH, Hansen LS, Pedersen M, Dejgaard T, Hansen J, Hall GV, Thomsen C, Solomon TP, Pedersen BK, Krogh-Madsen R. Changes in insulin sensitivity precede changes in body composition during 14 days of step reduction combined with overfeeding in healthy young men. J Appl Physiol (1985). 2012 Jul;113(1):7-15. doi: 10.1152/japplphysiol.00189.2011. Epub 2012 May 3. PMID 22556394